CLINICAL TRIAL: NCT00294931
Title: A Phase II Trial of Irinotecan, Carboplatin, Bevacizumab in the Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Irinotecan, Carboplatin, Bevacizumab in the Treatment of Patients With Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 90; AVF3256s
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-01

CONDITIONS: Carcinoma, Small Cell Lung
Keywords: Lung Cancer, Small Cell; Extensive
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Carboplatin; Bevacizumab

INTERVENTIONS:
Drug: irinotecan
Drug: carboplatin
Drug: bevacizumab

SUMMARY:
This multicenter phase II trial is designed to study the unique combination of chemotherapy (irinotecan./carboplatin) and bevacizumab in the extensive-stage setting. This clinical setting seems ideal for evaluation of the role of bevacizumab in delaying progression and prolonging survival.

DETAILED DESCRIPTION:
Eligible patients will receive 6 courses of irinotecan, carboplatin, and bevacizumab. The interval between chemotherapy courses will be 28 days. If after 6 courses of treatment, patient's response is a CR/PR/SD they will continue on Bevacizumab until tumor progression or up to 6 cycles (6 months) total.

Treatment sequence:

* Irinotecan 60mg/m2 on days 1, 8, and 15
* Carboplatin AUC=4 day 1 only
* Bevacizumab 10 mg/kg days 1 and 15

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed small cell lung cancer,extensive stage disease.
* Measurable or evaluable disease
* No previous chemotherapy
* Able to perform activities of daily living with minimal assistance
* Adequate hematological, live and kidney function
* Provide written informed consent

Exclusion Criteria:

* Limited stage disease
* PEG or G tubes
* Hemoptysis
* Abdominal fistula, perforation, or abscess within the previous 6 months
* Women who are pregnant or lactating
* Proteinuria
* Serious nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled or serious cardiovascular disease
* Uncontrolled brain metastasis
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days; Fine needle aspiration within 7 days
* Patients requiring full-dose anticoagulation must be on a stable dosing schedule prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
median time to progression

SECONDARY OUTCOMES:
overall toxicity
overall response rate
duration of response
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (4):
- United States (4):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Greco FA, Zubkus JD, Murphy PB, Saez RA, Farley C, Yardley DA, Burris HA 3rd, Hainsworth JD. Phase II trial of irinotecan, carboplatin, and bevacizumab in the treatment of patients with extensive-stage small-cell lung cancer. J Thorac Oncol. 2009 Dec;4(12):1555-60. doi: 10.1097/JTO.0b013e3181bbc540. PMID 19875975
- See also: Published article in the Journal of Thoracic Oncology — http://journals.lww.com/jto/pages/articleviewer.aspx?year=2009&issue=12000&article=00018&type=abstract